CLINICAL TRIAL: NCT01326494
Title: Reducing the Acute Care Burden of Childhood Asthma on Health Services in British Columbia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Bruce Carleton, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H10-00184
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Upper Respiratory Tract Infection; Asthma
Keywords: Upper Respiratory Tract Infection; Asthma; URTI induced exacerbation of Asthma
MeSH Terms: conditions — Respiratory Tract Infections; Asthma | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Oral Cortico Steroid (Active Comparator): A filled prescription will be given to be used upon early onset of symptoms.
  Interventions: Drug: Arm 1 Oral Cortico Steroids
- Usual care for Asthma treatment (No Intervention): monitor the readmission of URTI induced asthma in children over a 12 month period

INTERVENTIONS:
Drug: Arm 1 Oral Cortico Steroids — Prednisolone: 1 mg / kg per day course of dose for 5 days up to child's weight of 20 kgs.
  Dexamethasone: 0.3mg/kg per dose for 3 days (minimum weight 20 kgs )
  Other Names: Prednisone
  Arms: Arm 1 Oral Cortico Steroid

SUMMARY:
The purpose of this study is to investigate the benefits of giving filled prescription of a medication to be used upon early onset of symptoms of URTI induced asthma. The hope is to reduce the need to present to Health Care centres for treatment.

DETAILED DESCRIPTION:
In Canada, asthma affects more the 12% of children. Exacerbation are a common feature of asthma. In children, upper respiratory tract infection (URTI's) are responsible for over 80% of asthma exacerbation.

Experts in asthma care acknowledge this critical problem and have developed guidelines to reduce asthma exacerbation.

The criteria for participation in this study to have 2 or more presentations to a Health Service centre in the past 12 months for URTI induced asthma. These patients will be followed and interviewed monthly over a 12 month period to investigate whether the use of Oral cortico-steroids upon early onset of URTI induced asthma prevents the need for presentation to hospital

ELIGIBILITY:
Inclusion Criteria:

* 2 or more presentations to Emergency department in a 12 month period

Exclusion Criteria:

* less then 2 presentations to Emergency department in a 12 month period

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Reduction of representation to Health Services for Exacerbation of URTI induced asthma | One year
  To review the effect of medication given at early onset of symptoms have on reducing the presentation to Health Services and Emergency Departments.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Carleton, B.Pharm, Pharm.D., Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada